CLINICAL TRIAL: NCT05349851
Title: Clinical Registry of Adverse Effects in the Preparation for Colonoscopy in Patients With Advanced Renal Failure
Brief Title: Bowel Cleansing With Renal Impairment
Acronym: BC-RIMP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Marco Antonio Alvarez Gonzalez (Other)
Collaborators: Complejo Hospitalario de Navarra (Other); Althaia Xarxa Assistencial Universitària de Manresa (Other)
Responsible Party: Sponsor-Investigator, Marco Antonio Alvarez Gonzalez, Principal Investigator, Parc de Salut Mar
Organization: Parc de Salut Mar (Other)
Other Study IDs: 2020/9515
Record Dates: First submitted 2022-03-31; First posted 2022-04-27 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Renal Impairment; Adverse Effects of Medical Drugs
Keywords: Colonoscopy; Bowel cleansing; Renal impairment; Hydroelectrolytic adverse effects
MeSH Terms: conditions — Renal Insufficiency | interventions — Blood Specimen Collection; Urinalysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Renal failure patiens: Patients with advanced renal failure
  Interventions: Other: Follow-up with blood and urine analysis

INTERVENTIONS:
Other: Follow-up with blood and urine analysis — The patients will receive the preparation standards according to the usual clinical practice of each center. On the day of the colonoscopy, patient will be informed about this study and the informed consent will be requested to record the study information. Then, an analysis will be carried out. A second visit will be carried out, follow-up at 3-7 days, which will include a clinical interview and an analysis, being the unique intervention that patients receive.

SUMMARY:
Bowel preparation for colonoscopy requires the administration of large amounts of fluids that can cause fluid and electrolyte disturbances and volume overload, especially in patients with advanced renal failure. Polyethylene glycol-based regimens are considered safe, even in patients with advanced renal failure. However, the incidence of adverse effects (AEs) in routine clinical practice is unknown. The main objective of this study is to carry out a prospective, observational, multicenter clinical registry of renal AE of the preparation for colonoscopy, in patients with advanced renal failure, within the usual clinical practice of the preparation. Variables related to kidney function, bowel-cleansing efficacy, and tolerance will also be recorded. A segmented analysis will be performed in patients with substitutive renal therapy (hemodialysis or peritoneal dialysis).

DETAILED DESCRIPTION:
Introduction: Bowel preparation for colonoscopy requires the administration of large amounts of fluids that can cause fluid and electrolyte alterations and volume overload, especially in patients with advanced renal failure. Routine clinical practice of bowel preparation with polyethylene glycol-based regimens, including in patients with advanced renal failure, is considered safe. The hydroelectrolytic AEs and worsening of renal failure are generally mild and transient. However, the incidence of AEs in routine clinical practice is unknown, because there is no prospective record of the incidence of renal AEs in these patients.

Objectives:

1. Principal. To carry out a clinical registry of the renal AEs of the preparation for colonoscopy, in patients with advanced renal failure, within the usual clinical practice of the preparation.
2. Secondary:

   * Study the efficacy of intestinal cleansing using the Boston bowel preparation scale.
   * Study the patient-reported experience measures (PREMs) in terms of tolerability and acceptance of bowel preparation.

Study of the population and sample size: Outpatients with a scheduled colonoscopy for any indication and with moderate or severe renal impairment. Ages: 18-80, excluding partial colectomy, severe constipation, active intestinal disease, severe heart or liver failure, pregnancy or lactation, and refusal to authorize the clinical record of information. We calculated a sample size of 237 subjects to show an incidence of renal AD of 10%, with a precision of 4%.

Methods: Identify patients with a scheduled colonoscopy who present advanced renal failure, in the 60 days prior to the colonoscopy. Carry out a prospective, observational, multicenter clinical registry of the routine clinical practice of preparation for colonoscopy. Variables related to renal function, the efficacy of intestinal cleansing, and tolerance will be recorded. A segmented analysis will be performed in patients with substitutive renal therapy (hemodialysis or peritoneal dialysis). The data will be collected on the REDCap-AEG online platform, which can be accessed by researchers from each center through an identification code, respecting the current Organic Law on Data Protection.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients or hospitalized patients with previously scheduled colonoscopy with any indication: screening, follow-up or symptoms.
* Diagnosis of stage 3B-5D chronic renal failure (creatinine clearance less than 45 ml / min / 1.73 m2).

Exclusion Criteria:

* Age less than 18 years or greater than 80 years
* Partial or total colectomy
* Severe constipation
* Active inflammatory bowel disease
* Severe hepatic impairment (Child Pugh Classification C)
* Pregnancy or breastfeeding
* Refusal to authorize the clinical registration of the information

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatients with a scheduled colonoscopy for any indication and with moderate or severe renal impairment
Sampling Method: Non-Probability Sample
Enrollment: 237 (Estimated)
Dates: Start 2021-10-05 (Actual); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Global incidence of renal adverse effects (AEs) | 3 hours to 7 days after laxative intake
  Global incidence of renal adverse effects (AEs) (yes/no) if any of the following variables have an abnormal value in serum: sodium, potassium, calcium, chloride, bicarbonate, creatinine, or the glomerular filtrate rate calculated with the MDRD formula and the CKD-EPI formula.

SECONDARY OUTCOMES:
Serum sodium concentration | 3 hours to 7 days after laxative intake
  Any abnormal value in serum sodium concentration.
Serum potasium concentration | 3 hours to 7 days after laxative intake
  Any abnormal value in serum potasium concentration.
Serum ionized calcium concentration | 3 hours to 7 days after laxative intake
  Any abnormal value in serum ionized calcium concentration.
Serum chloride concentration | 3 hours to 7 days after laxative intake
  Any abnormal value in serum chloride concentration.
Serum bicarbonate concentration | 3 hours to 7 days after laxative intake
  Any abnormal value in serum bicarbonate concentration.
Serum creatinine concentration | 3 hours to 7 days after laxative intake
  Any abnormal value in serum creatinine concentration.
Glomerular filtration rate | 3 hours to 7 days after laxative intake
  Glomerular filtration rate calculated with the MDRD formula and the CKD-EPI formula.
Serum phosphorus concentration | 3 hours to 7 days after laxative intake
  Any abnormal value in serum phosphorus concentration.
Serum magnesium concentration | 3 hours to 7 days after laxative intake
  Any abnormal value in serum magnesium concentration.
Blood pH | 3 hours to 7 days after laxative intake
  Blood pH measurement
Hemoglobin concentration | 3 hours to 7 days after laxative intake
  Mean corpuscular hemoglobin
Blood platelets | 3 hours to 7 days after laxative intake
  Number of blood platelets
Adequate bowel cleansing for colonoscopy | At the moment of colonoscopy
  Application of the Boston Bowel Preparation Scale to evaluate colonoscopy bowel cleansing. The efficacy of bowel preparation will be rated by blinded endoscopists using the Boston Bowel Preparation Scale (BBPS). Adequate bowel cleansing will be defined as a BBPS of 2 or more points in every segment of the colon and inadequate bowel cleansing will be defined by at least one of the colon segments with less than 2 points.
Adhrence to laxative intake | 3-5 hours after laxative intake (at the colonoscopy appointment)
  Adhrence to laxative intake recorded as >75% of the quantity of laxative intake reported in a questionarie administered with the help of an investigator.
Time from last intake of laxative to the colonoscopy | 3-5 hours after laxative intake (at the colonoscopy appointment)
  Interval in hours between last intake of laxative and the colonoscopy.
Patient-reported experience measures (PREMs) questionnaire of laxative intake | 3-5 hours after laxative intake (at the colonoscopy appointment)
  Patient-reported experience measures (PREMs) questionnaire of laxative intake, administered with the help of an investigator. Descriptive subjective scale: Very bad, bad, average, good, very Good.
Early side effects of laxative intake | 3-5 hours after laxative intake (at the colonoscopy appointment)
  Early side effects of laxative intake. Structured questionnaire nausea, vomiting, dizziness, thirst, headache, abdominal bloating. Non structured for other side effects.
Late side effects of laxative intake | 3-7 days after laxative intake
  Structured questionnaire nausea, vomiting, dizziness, thirst, headache, abdominal bloating, abdominal pain, mental confusion, asthenia, dyspnea, peripheral edema. Non structured for other side effects.
Need of urgent consultation | 3 hours to 7 days after laxative intake
  Number of participants requiring medical consultation for kidney related problems, including emergency room or nephrologist consultation.
Need for hospital admission | 3 hours to 7 days after laxative intake
  Number of participants requiring hospital admission for any kidney related causes.
Need of any drug treatment, new treatment or modification, that may affect kidney function or serum electrolytes | 3 hours to 7 days after laxative intake
  Number of participants that require outpatient medication change after the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Marco A Álvarez, MD, PhD, Principal Investigator — Althaia Xarxa Assistencial Universitària de Manresa; Institut Hospital del Mar d'investigacions mèdiques, Barcelona.; Eduardo Albéniz, MD, PhD, Principal Investigator — Hospital Universitario de Navarra; Navarrabiomed; UPNA; IdiSNA
Locations (2):
- Spain (2):
  - Althaia Xarxa Assistencial Universitària de Manresa, Manresa, Catalonia
  - Hospital Reina Sofía, Tudela, Navarre

IPD SHARING:
Plan to Share IPD: No